CLINICAL TRIAL: NCT01840644
Title: Validity and Reliability of Perceived Exertion Rating Scale in Children With Traumatic Brain Injury, Cerebral Palsy and Typically Developed
Brief Title: Validity and Reliability of Perceived Exertion Rating Scale in Children With Brain Damage
Status: Completed | Type: Observational
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 920090351
Record Dates: First submitted 2010-02-15; First posted 2013-04-26 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Traumatic Brain Injury; Cerebral Palsy
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Palsy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all participants: Walking on treadmill, different velocities and incline
  Interventions: Other: Walking on treadmill, different velocities and incline

INTERVENTIONS:
Other: Walking on treadmill, different velocities and incline — Walking on treadmill twice, with one week interval in each session the child will walk in different velocities and incline
  Other Names: RPE

SUMMARY:
The purpose of this study is to examine the reliability and validity of the rating of perceived exertion scale in children post severe traumatic brain injury during treadmill exercise.

DETAILED DESCRIPTION:
walking on a treadmill twice- one weeks interval five intensity level in each session

ELIGIBILITY:
Inclusion Criteria:

* Children post severe closed head injury (Glasgow Coma Scale [GCS] score at admission to emergency room of ≤8, at least one year post trauma
* Ages 7 to 12 years
* (3) independent ambulation (foot orthoses permitted).
* Children with Cerebral palsy, GMFCS 1 or 2, ages 7 to 12 years. Typically developed controls.

Exclusion criteria:

* Cannot understand simple instructions

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children post severe TBI Children with CP TD control
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
OMNI scale, a pictorial perceived extortion scale for children | three meetings once a week.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Katz, Phd, Study Director — Alyn rehabilitation center
Locations (1):
- Alyn Children's Rehabilitation Hospital, Jerusalem, Israel